CLINICAL TRIAL: NCT03908593
Title: Evaluation of the Efficacy of Different Duration of a Proton Pump Inhibitor in the Prevention of Upper Gastrointestinal Mucosal Injury in Patients Taking 12-month Dual Antiplatelet Therapy After Coronary Artery Bypass Grafting
Brief Title: Proton Pump Inhibitor Preventing Upper Gastrointestinal Injury In Patients On Dual Antiplatelet Therapy After CABG
Acronym: DACAB-GI-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Lifen YU, Associate Professor, Department of Gastroenterology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IISR-2016-101603 (RJ)
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Gastrointestinal Ulcer (Peptic) or Erosion; Anti-Platelet Therapy; Coronary Artery Bypass
Keywords: Gastrointestinal; Mucosal injury; Antiplatelet; Coronary artery bypass grafting; Prevention
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One month of therapy (Active Comparator): Pantoprazole, 40mg, tablet, oral, once daily for 1 month
  Interventions: Drug: Pantoprazole
- Twelve months of therapy (Experimental): Pantoprazole, 40mg, tablet, oral, once daily for 12 months
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Pantoprazole (40mg qd) will be concomitant used with DAPT
  Other Names: PANTOLOC, Tablet from Takeda Pharmaceutical Company Limited

SUMMARY:
The purpose of this study is to compare the efficacy and safety for 12- vs. 1-month of pantoprazole treatment in preventing dual antiplatelet therapy (DAPT)-related upper gastrointestinal mucosal injury after coronary artery bypass grafting (CABG).

To date, there has been no study using esophagogastroduodenoscopy (EGD) to compare the differences in upper gastrointestinal mucosal injury (including reflux esophagitis) after 6 and 12 months of PPI treatment combined with two different DAPT regimens (clopidogrel plus aspirin or ticagrelor plus aspirin).

DETAILED DESCRIPTION:
This prospective trial was designed as a single-center, open-label, randomized controlled trial with patients allocated in a ratio of 1:1. Within 3 days after CABG, patients willing to participate in the study will be carefully evaluated by a cardiac surgeon together with a gastroenterologist based on inclusion and exclusion criteria. Patients will be followed up to 12 months post-randomization unless death. The outcome will be collected at 2±1 days, 9±2 days, 1 month, 3 months (phone call), 6 months, 9 months (phone call), and 12 months after CABG surgery, respectively. 13C urea breath testing is used to detect Helicobacter pylori (H. pylori) infection before enrollment. At 6 and 12 months post-randomization, routine laboratory tests and EGD will be performed respectively. Computed tomographic angiography (CTA) or coronary angiography (CAG) is also required at 12 months post-randomization.

Definition of end of the study

1. The date on which the last subject completed the last follow-up was the endpoint of this study.
2. During the follow-up period, if the patient's biopsy pathological report showed that EGD detects precancerous lesions (e.g., atypical hyperplasia, low-grade or high-grade internal neoplasia, etc.) or malignant lesions.
3. Patients randomized to the control group (1-month pantoprazole treatment group) should continue PPI treatment if GERD-Q questionnaire score 8, endoscopic findings of reflux esophagitis (LA-A and above), gastroduodenal mucosal injury of modified Lanza score of 4, or upper gastrointestinal bleeding at any time during the follow-up period.

Following the ITT principle, all patients randomized in this study should be evaluated for primary and secondary endpoints regardless of changes in PPI treatment. Thus, patients in the 1-month pantoprazole treatment group required PPI treatment at any time after 1 month and could also be assessed for primary and secondary endpoints.

According to the results of the preliminary study, the cumulative incidence rate of severe gastric and duodenal bulb erosion and ulcers of the 1-month PPI treatment group is assumed to be 36%, and that of the 12-month PPI treatment group was assumed to be 18%. Based on a two-sided α of 0.05 and a randomization ratio of 1:1, a total of 186 subjects are required to provide a power of 80%. Considering a 20% drop-out rate, the sample size of 232 subjects was determined.

In this study, all subjects received pantoprazole treatment for at least 1 month after CABG. Due to the COVID-19 pandemic, some subjects are unable to return to the center for study drugs and/or follow-up 1 month after the randomization. Those subjects who are unable to receive subsequent randomization intervention, will be excluded from the modified full analysis set and not included in the effectiveness analysis. Considering the statistical power of the study, randomized subjects will be added until the effective randomized intervention number reaches the predetermined sample size.

Two subgroup analyses will be performed in this study, including (1) H. pylori infection: negative and positive; (2) DAPT: aspirin + clopidogrel and aspirin + ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

Each patient should meet all of the inclusion criteria and none of the exclusion criteria for this study:

1. Provision of signed informed consent prior to any study specific procedures.
2. Male or female, age ≥ 18 years at the time of consent.
3. Planned or initiated use of 12 months of DAPT (aspirin plus clopidogrel or aspirin plus ticagrelor) immediately following primary isolated elective CABG surgery.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled.

1. History of previous active peptic ulcer within 3 months prior to enrollment.
2. Planned use of PPIs to treat acid-associated disorders (e.g. gastroesophageal reflux disease, GERD)
3. Contraindications for aspirin, clopidogrel, ticagrelor and pantoprazole use (e.g. known allergy)
4. Anticipated concomitant oral or intravenous therapy with strong cytochrome P450 3A4 (CYP3A4) inhibitors or CYP3A4 substrates with narrow therapeutic indices, that cannot be stopped for the course of the study.

   * Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir
   * CYP3A4 substrates with narrow therapeutic index: quinidine, simvastatin at doses > 40mg daily or lovastatin at doses > 40mg daily.
5. Need for chronic oral anticoagulant therapy or chronic low-molecular-weight heparin.
6. Women of child-bearing potential who are not willing to use a medically accepted method of contraception that is considered reliable in the judgement of investigator OR women who have a positive pregnancy test at enrollment or randomization OR women who are breasting-feeding.
7. Inability of patient to understand and/or comply with study procedures and/or follow up, in the opinion of the investigator, OR any conditions that, in the opinion of the investigator, many render the patient unable to complete the study.
8. Any condition outside the atherothrombotic study area with a life expectancy of less than 1 year.
9. Participation in another clinical study with an investigational product within 28 days prior to enrolment or previous randomization to an investigational product in another ongoing clinical study.
10. Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study (eg, long-term concomitant treatment with non-steroidal anti-inflammatory drugs [NSAIDs])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with gastroduodenal erosions and ulcers evaluated by EGD. | within 12 months after randomization
  Gastroduodenal erosions and ulcers will be assessed according to the Lanza Endoscopic Scoring System. Lanza score is a categorical score (0-4) and defined as follows: 0, normal; 1, mucosal hemorrhages only; 2, 1-2 erosions; 3, 3-10 erosions; 4, >10 erosions or an ulcer ≥3 mm. In addition, ≥1 ulcer with a diameter no less than 5mm will be grouped separately.

SECONDARY OUTCOMES:
Percentage of patients with gastroduodenal erosions and ulcers evaluated by EGD. | 6 months after randomization
  Gastroduodenal erosions and ulcers will be assessed according to the Lanza Endoscopic Scoring System (0-4). In addition, ≥1 ulcer with a diameter ≥5mm will be grouped separately.
Cumulative rate of patients with upper gastrointestinal bleeding (UGIB) according to the modified TIMI criteria. | within 12 months after randomization
  According to the definition of non-CABG related bleeding in the modified TIMI criteria, the severity of UGIB is classified into 3 grades: major, minor and minimal. 1, Major: Clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥5 g/dL. 2, Minor: Clinically overt signs of UGIB, resulting in hemoglobin drop of 3 to <5 g/dL. 3, Minimal: Any overt bleeding event that does not meet the criteria above. According to the consensus updated by the Asia-Pacific working group in 2018, patients with hemodynamic shock and signs of UGIB should be offered urgent endoscopy after resuscitation and stabilization (Gut 2018; 67:1757-68).
Percentage of patients with reflux esophagitis evaluated by EGD. | 12 months after randomization
  According to the Los Angeles classification, endoscopic reflux esophagitis was assigned a grade from A to D.
Percentage of patients with reflux esophagitis evaluated by EGD. | 6 months after randomization
  According to the Los Angeles classification, endoscopic reflux esophagitis was assigned a grade from A to D.

OTHER OUTCOMES:
Cumulative rate of patients with major adverse cardiovascular events (MACE). | up to 12 months
  MACE: composite of cardiovascular death, myocardial infarctions, or stroke.
The failure rate of grafts assessed by computed tomographic angiography or coronary angiography. | up to 12 months
  Graft failure was assessed according to the modified Fitzgibbon classification: Stenosis ≥50% or occlusion of the graft or distal anastomosis (type B or O)
Cumulative rate of patients with all-cause death | up to 12 months
  All-cause death: Death from all causes during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lifen Yu, MD, Ph.D, Principal Investigator — Department of Gastroenterology, Ruijin Hospital; Qiang Zhao, MD, Ph.D, Principal Investigator — Department of Cardiovascular Surgery, Ruijin Hospital; Yunpeng Zhu, MD, Study Director — Department of Cardiovascular Surgery, Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu Y, Wang X, Yang Y, Liu L, Zhao Q, Yu L. Proton pump inhibitor in the prevention of upper gastrointestinal mucosal injury associated with dual antiplatelet therapy after coronary artery bypass grafting (DACAB-GI-2): study protocol for a randomized controlled trial. Trials. 2022 Jul 15;23(1):569. doi: 10.1186/s13063-022-06464-w. PMID 35840999